CLINICAL TRIAL: NCT05889390
Title: [A Prospective, Randomized Trial to Assess the Added Value of Concomitant Modulated Electro-hyperthermia in Breast Cancer Patients Receiving Neoadjuvant Chemotherapy - an Investigator Initiated Study]
Brief Title: Neoadjuvant Concomitant Modulated Electro-hyperthermia in HER2-negative Breast Cancer
Acronym: NeoHTerMa
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Marcell Szasz, Dr. A. Marcell Szasz, PhD, Head of Research at the Department of Internal Medicine and Oncology, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeoHTerMa
Record Dates: First submitted 2023-03-03; First posted 2023-06-05 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: HER2-negative Breast Cancer
Keywords: hyperthermia; modulated electro-hyperthermia; oncothermia; breast cancer
MeSH Terms: conditions — Hyperthermia; Breast Neoplasms | interventions — Paclitaxel; Carboplatin; AC protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- wTAX (+ carboplatin) +AC (Active Comparator): 1. wTAX: Weekly paclitaxel (+ carboplatin in the case of triple-negative breast cancer) for 12 weeks
  2. AC: Doxorubicin/Cyclophosphamide every three-weeks, 4x
  3. Breast cancer tumor removal surgery (if feasible)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Cyclophosphamide/Doxorubicin; Procedure: Breast cancer removal surgery
- wTAX (+ carboplatin) +AC + mEHT (Experimental): 1. wTAX + mWEHT
     1. wTAX: Weekly paclitaxel (+ carboplatin in the case of triple-negative breast cancer) for 12 weeks
     2. mEHT: Concomitant modulated electro-hyperthermia using the Oncotherm EHY-2030 device, 3 times per week, for 12 weeks
  2. AC: Doxorubicin/Cyclophosphamide every three-weeks, 4x
  3. Breast cancer tumor removal surgery (if feasible)
  Interventions: Device: Oncotherm EHY-2030; Drug: Paclitaxel; Drug: Carboplatin; Drug: Cyclophosphamide/Doxorubicin; Procedure: Breast cancer removal surgery

INTERVENTIONS:
Device: Oncotherm EHY-2030 — Oncotherm EHY-2030 is a non-invasive electromagnetic devices with known anti-tumoral effects. It operates in a precision capacitive coupled impedance matched way, working on a radiofrequency of 13.56 MHz. mEHT exploits various biophysical differences of cancer cells. For example, energy absorption on the membrane rafts is different than those of healthy host cells, and damage-associated molecular patterns (DAMPS) will also occur leading to programmed or immunogenic tumor cell death. mEHT can enhance DNA fragmentation of tumor cells, increase the fraction of cells with low mitochondrial membrane potential, increase the concentration of intracellular Ca2+, increase the Fas, c-Jun N-terminal kinases and MAPK/ERK signaling pathways, increase the expression of pro-apoptotic Bcl-2 family proteins and can up-regulate the expression of genes associated with the molecular function of cell death (EGR1, JUN, and CDKN1A) and silencing others associated with cytoprotective functions.
  Arms: wTAX (+ carboplatin) +AC + mEHT
Drug: Paclitaxel — weekly paclitaxel for 12 weeks
Drug: Carboplatin — added to weekly paclitaxel if patient has triple-negative breast cancer
Drug: Cyclophosphamide/Doxorubicin — according to the AC protocol
Procedure: Breast cancer removal surgery — Either breast-conserving surgery or total mastectomy after the neoadjuvant chemotherapy with or without mEHT (if feasible)

SUMMARY:
The aim of this study is to investigate whether the application of concomitant modulated electro-hyperthermia in a neoadjuvant chemotherapeutic setting is beneficial for patients with HER2-negative, stage II-III breast cancer.

DETAILED DESCRIPTION:
This study is a pivotal, randomized (1:1), open-label, two-treatment group, single-centre trial of Oncotherm EHY-2030, a modulated electro-hyperthermia (mEHT) device. Female patients aged 18 years or older with locally advanced, unilaterally localized HER2-negative breast cancer requiring neoadjuvant treatment are eligible for the study.

In the study, the wTAX (+ carboplatin) +AC neoadjuvant chemotherapy protocol will be administered according to the routine daily regimen, with or without mEHT three times a week during the wTAX (+ carboplatin) period. Carboplatin will be administered for patients with triple-negative breast cancer only.

Primary objective: to compare whether the percentage of tumor size decrease determined by imaging techniques is different in the two treatment groups?

Secondary and other objectives:

* Is complete pathological response (pCR) more common in the mEHT-treated group?
* Does the pattern of treatment response (pCR : pPR : pNR) differ between the two groups?
* Is the quality of life of patients different in the two study groups?
* Is there any treatment-related changes in the routine laboratory parameters such as blood count, liver enzymes, renal function? And do these differ in the two study arms?
* Safety and tolerability analysis of the device.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Female patient
3. Life expectancy ≥ 6 months
4. De novo histological/cytological diagnosis of HER2-negative (triple-negative or ER/PR+) breast tumor involving one breast
5. Diagnosis of breast tumor ≤ 40 days
6. Locally advanced stage disease (stage II and III) requiring neoadjuvant treatment - according to the following criteria:

   1. Primary breast tumor ≥ 20 mm in size and/or
   2. Presence of axillary lymph node metastases
   3. Optimal surgical intervention without neoadjuvant chemotherapy is not feasible
7. ECOG status: 0-2
8. Suitable for and designated by the investigator for neoadjuvant therapy with wTAX + (carboplatin) + AC chemotherapeutic agent
9. Willingness to participate in the trial and signed the informed consent form for the protocol

Exclusion Criteria:

1. Patient is ≤ 18 years of age.
2. Tumor of both breasts.
3. Diagnosis of breast tumor > 40 days
4. HER2 positive breast tumor
5. Has already received some anticancer therapy
6. Any previous cancer requiring anti-tumor treatment within 5 years prior to selection, except: in situ cervical or uterine cancer and non-melanoma skin cancer.
7. Co-existing serious diseases:

   1. Presence of severe neuropathy requiring medical treatment, diabetic neuropathy.
   2. Clinically significant hematological, hepatic or renal dysfunction, as defined below:

      * Neutrophil count < 1.5 G/L and platelet count < 100 G/L
      * bilirubin > 1.5 times the upper limit of normal range (ULN), except for known Gilbert's disease
      * AST and/or ALT > 2.5 times the upper limit of the normal range
      * Serum creatinine > 1.5 times the upper limit of the normal range.
   3. Clinically significant cardiovascular disease in the medical history, unless the disease is adequately controlled. E.g. New York Heart Association (NYHA) Class II or worse congestive heart failure (moderate limitation of physical activity; well-being at rest but normal activity is associated with fatigue, rapid heart rate or dyspnoea).
   4. Uncontrolled hypertension with resting systolic ≥ 180 mmHg, resting diastolic ≥ 110 mmHg.
   5. Resting sinus tachycardia with a pulse ≥ 110/min.
   6. History of sympathetic or treatment-naive cardiac arrhythmia. Atrial fibrillation or flutter controlled with medication is not an exclusion for participation in the study.
   7. Major cardiovascular event (e.g. myocardial infarction, unstable angina, cerebral vascular accident (CVA), etc.) in the 6 months prior to randomisation.
   8. Active infection or severe underlying disease that renders the patient unfit for treatment according to the study protocol.

      * A current diagnosis of chronic hepatitis, Hepatitis B surface antigen positive, Hepatitis C antibody positive and/or other clinically active liver disease requiring treatment.
      * Known HIV infection.
      * Untreated thyroid disease.
      * Systemic autoimmune disease.
   9. Any psychiatric condition in the medical history that may result in the patient being unable to understand or comply with the requirements of the study, having reduced communication skills or being unable to give informed consent.
8. Need for concomitant anti-tumor therapy in addition to wTAX + (carboplatin) + AC protocol
9. Any active medical device implanted in the anatomical area, such as pacemakers.
10. Known severe hypersensitivity to any of the chemotherapies used in the study.
11. Pregnancy or breast-feeding (patients of childbearing potential must use effective contraception throughout the study and for 3 months after the end of treatment). The method of effective contraception is at the discretion of the investigator.
12. History of drug or alcohol dependence within 6 months prior to screening.
13. Unable to comply with the study plan for medical, psychological, family, geographical or other reasons.
14. Institutionalisation by administrative or judicial decision.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Residual size of the primary tumor, determined by imaging techniques (in percentage) | change from baseline at 6 months
  Using breast MR measurements, the the residual size of the primary tumor will be specified for all patients (in percentage). The comparison of these between the two study arms will serve as the primary outcome measure.
  Calculation: The tumor size after the 6-months treatment period (in mm) will be divided by the size measured prior treatment (in mm). The quotient will be given as a percentage and subtracted from 100.

SECONDARY OUTCOMES:
Percentage of complete pathological response | 9 months
  Comparison of the percentage of complete pathological responses between the two groups
Treatment response patterns | 9 months
  Comparison of the pathological response categories (pCR : pPR : pNR) between the two groups
Comparison of surgical procedure ratios | 9 months
  It will be compared whether the ratio of two main breast surgery types (breast-conserving surgery vs. total mastectomy) differ between the two study arms.
Effect of treatment on white blood cell counts | through study completion, an average of ~8 months
  White blood cell counts (in G/L) will be measeured at every patient visit, and their longitudinal change will be analyzed using mixed-effect statistical modeling techniques.
Effect of treatment on red blood cell counts | through study completion, an average of ~8 months
  Red blood cell counts (in T/L) will be measeured at every patient visit, and their longitudinal change will be analyzed using mixed-effect statistical modeling techniques.
Effect of treatment on platelet counts | through study completion, an average of ~8 months
  Platelet counts (in G/L) will be measeured at every patient visit, and their longitudinal change will be analyzed using mixed-effect statistical modeling techniques.
Effect of treatment on hemoglobin levels | through study completion, an average of ~8 months
  Hemoglobin level of patients (in g/L) will be measeured at every patient visit, and their longitudinal change will be analyzed using mixed-effect statistical modeling techniques.
Effect of treatment on hematocrit levels | through study completion, an average of ~8 months
  Hematocrit level of patients (in L/L) will be measeured at every patient visit, and their longitudinal change will be analyzed using mixed-effect statistical modeling techniques.
Number of treatments where the planned power output of the Oncotherm EHY-2030 device could not be reached | 3 months
  For an optimal treatment, the Oncotherm EHY-2030 device must reach its maximum output for 30 minutes. The number of treatments where this optimal outpur could not be reached will be reported.
Longitudinal analysis of the EORTC QLQ-C30 questionnaire's total scores | through study completion, an average of ~8 months
  The European Organisation for Research and Treatment of Cancer 30-item quality of life questionnaire for cancer patients (EORTC QLQ-C30) total scores will be calculated as per the official quidelines, and their longitudinal change will be analyzed using mixed-effect statistical modeling techniques.
  Scoring of the questionnaire will be performed as per the official instructions of EORTC
Longitudinal analysis of the EORTC QLQ-BR23 questionnaire's total scores | through study completion, an average of ~8 months
  The European Organisation for Research and Treatment of Cancer 23-item quality of life questionnaire for breast cancer patients (EORTC QLQ-BR23) total scores will be calculated as per the official quidelines, and their longitudinal change will be analyzed using mixed-effect statistical modeling techniques.
  Scoring of the questionnaire will be performed as per the official instructions of EORTC
Longitudinal analysis of the EQ-5D-5L questionnaire scores | through study completion, an average of ~8 months
  The questionnaire will be assessed as per official guidelines.
  EuroQol's 5-dimension health-related quality of life instrument (EQ-5D-5L) questionnaire scores' longitudinal change will be analyzed using mixed-effect statistical modeling techniques.
  Scoring of the questionnaire will be performed as per the official instructions of EuroQol.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. | through study completion, an average of ~8 months
  All adverse events will be assessed and classified by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
  Using descriptive statistics, the number of occurrances will be listed for both study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Magdolna Dank, M.D./Ph.D., Principal Investigator — Semmelweis University
Locations (1):
- Division of Oncology, Department of Internal Medicine and Oncology, Semmelweis University, Budapest, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szasz AM, Minnaar CA, Szentmartoni G, Szigeti GP, Dank M. Review of the Clinical Evidences of Modulated Electro-Hyperthermia (mEHT) Method: An Update for the Practicing Oncologist. Front Oncol. 2019 Nov 1;9:1012. doi: 10.3389/fonc.2019.01012. eCollection 2019. PMID 31737558
- [Background] Herold Z, Szasz AM, Dank M. Evidence based tools to improve efficiency of currently administered oncotherapies for tumors of the hepatopancreatobiliary system. World J Gastrointest Oncol. 2021 Sep 15;13(9):1109-1120. doi: 10.4251/wjgo.v13.i9.1109. PMID 34616516
- [Background] Petenyi FG, Garay T, Muhl D, Izso B, Karaszi A, Borbenyi E, Herold M, Herold Z, Szasz AM, Dank M. Modulated Electro-Hyperthermic (mEHT) Treatment in the Therapy of Inoperable Pancreatic Cancer Patients-A Single-Center Case-Control Study. Diseases. 2021 Nov 3;9(4):81. doi: 10.3390/diseases9040081. PMID 34842668
- [Background] Szasz AM, Arrojo Alvarez EE, Fiorentini G, Herold M, Herold Z, Sarti D, Dank M. Meta-Analysis of Modulated Electro-Hyperthermia and Tumor Treating Fields in the Treatment of Glioblastomas. Cancers (Basel). 2023 Jan 31;15(3):880. doi: 10.3390/cancers15030880. PMID 36765840